CLINICAL TRIAL: NCT00480038
Title: WHODAS-II for Patients With Symptomatic Lumbar Disc Herniation
Brief Title: World Health Organization Disability Assessment Schedule (WHODAS-II) for Patients With Symptomatic Lumbar Disc Herniation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was so slow, that it made the study impossible. Organizational changes made it impossible for recruiting centers to continue recruitment
Sponsor: Kovacs Foundation (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FK-R-18
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Lumbar Disc Herniation
Keywords: symptomatic; lumbar disc herniation; disability; fear avoidance beliefs; quality of life
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule)
  Interventions: Other: WHODAS II

INTERVENTIONS:
Other: WHODAS II — To determine the measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule)

SUMMARY:
The main purpose of this study is to determine the measurement characteristics of WHODAS II (World Health Organization Disability Assessment Schedule), as well as to analyze its correlation with symptomatic lumbar disc herniation (Visual Analog Scale, VAS), disability (Spanish version of the Roland Morris Questionnaire, RMQ), fear avoidance beliefs and attitudes (Spanish version of the FAB Questionnaire, FABQ) and quality of life (SF-12). Measurements will be taken at baseline and 6 days later (day 7).

ELIGIBILITY:
Inclusion Criteria:

* Patients seen for symptomatic lumbar disc herniation
* Radiated pain concordant with nerve root
* With or without motor restriction
* Able to read and write
* Signed the informed consent form

Exclusion Criteria:

* Central nervous system pathology (with or without treatment)
* Diagnosis of rheumatic inflammatory disease or fibromyalgia
* Red flags for underlying systemic disease
* Criteria for diagnosis of symptomatic spinal stenosis
* Symptoms suggesting saddle anesthesia, cauda equina, loss of sphincter tone or paraparesis
* Motor deficit that progresses or does not improve in 6 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measurement characteristics of WHODAS-II | At baseline and at 7 days

SECONDARY OUTCOMES:
Correlation between WHODAS-II and VAS, RMQ, FABQ and SF-12 in symptomatic lumbar herniated disc | At baseline and at 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; José Luis Peña, MD, Principal Investigator — Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain
Locations (2):
- Spain (2):
  - Fundación Kovacs, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria

REFERENCES:
- [Background] Bombardier C. Outcome assessments in the evaluation of treatment of spinal disorders. Introduction. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3097-9. doi: 10.1097/00007632-200012150-00002. No abstract available. PMID 11124723
- [Background] Chwastiak LA, Von Korff M. Disability in depression and back pain: evaluation of the World Health Organization Disability Assessment Schedule (WHO DAS II) in a primary care setting. J Clin Epidemiol. 2003 Jun;56(6):507-14. doi: 10.1016/s0895-4356(03)00051-9. PMID 12873644
- [Background] van Tubergen A, Landewe R, Heuft-Dorenbosch L, Spoorenberg A, van der Heijde D, van der Tempel H, van der Linden S. Assessment of disability with the World Health Organisation Disability Assessment Schedule II in patients with ankylosing spondylitis. Ann Rheum Dis. 2003 Feb;62(2):140-5. doi: 10.1136/ard.62.2.140. PMID 12525383